CLINICAL TRIAL: NCT00359164
Title: A Randomized, Controlled, Double-Masked, Phase II Pilot Study of Visudyne® Photodynamic Therapy (PDT) (Low and Very Low Fluence) Combined With Bevacizumab (Avastin), in Patients With Subfoveal Choroidal Neovascularization (CNV) Secondary to Age Related Macular Degeneration (AMD)
Brief Title: Phase II Pilot Study of Visudyne® Photodynamic Therapy (PDT) (Low and Very Low Fluence) Combined With Bevacizumab.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Dr. Michael Potter, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C06-0202; V06-0157
Record Dates: First submitted 2006-07-28; First posted 2006-08-01 (Estimated); Last update posted 2008-08-14 (Estimated); Status verified 2008-08

CONDITIONS: Macular Degeneration
Keywords: AMD; Avastin; Visudyne; Medical condition being studied AMD
MeSH Terms: conditions — Macular Degeneration | interventions — Bevacizumab; Verteporfin; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- 1 (Active Comparator): Bevacizumab with verteporfin at Low Fluence Photodynamic Therapy.
  Interventions: Drug: Verteporfin Photodynamic Therapy (Low Fluence) and bevacizumab
- 2 (Active Comparator): Bevacizumab with verteporfin at Very Low Photodynamic Therapy.
  Interventions: Drug: Verteporfin Photodynamic Therapy (Very Low Fluence) and bevacizumab
- 3 (Sham Comparator): Bevacizumab with verteporfin with Sham Photodynamic Therapy.
  Interventions: Drug: Verteporfin Photodynamic Therapy (SHAM) and bevacizumab

INTERVENTIONS:
Drug: Verteporfin Photodynamic Therapy (Low Fluence) and bevacizumab — Bevacizumab 1.25 mg with verteporfin at Low Fluence (300 mW/cm2 delivered for 83 seconds [light dose of 25 J/cm2]) Photodynamic Therapy.
  Treatment at Baseline visit, followed by an "as needed" basis. Assessments monthly for bevacizumab and at 3-month intervals for combination therapy with verteporfin or sham.
  Other Names: Verteporfin = Visudyne; Bevacizumab = Avastin
  Arms: 1
Drug: Verteporfin Photodynamic Therapy (Very Low Fluence) and bevacizumab — Bevacizumab 1.25 mg with verteporfin at Low Fluence (150 mW/cm2 delivered for 83 seconds [light dose of 12.5 J/cm2]) Photodynamic Therapy.
  Treatment at Baseline visit, followed by an "as needed" basis. Assessments monthly for bevacizumab and at 3-month intervals for combination therapy with verteporfin or sham.
  Other Names: Verteporfin = Visudyne; Bevacizumab = Avastin
  Arms: 2
Drug: Verteporfin Photodynamic Therapy (SHAM) and bevacizumab — Bevacizumab with SHAM (150 mW/cm2 delivered for 83 seconds [light dose of 12.5 J/cm2]) Photodynamic Therapy.
  Treatment at Baseline visit, followed by an "as needed" basis. Assessments monthly for bevacizumab and at 3-month intervals for combination therapy with verteporfin or sham.
  Other Names: Verteporfin = Visudyne; Bevacizumab = Avastin
  Arms: 3

SUMMARY:
To determine if Visudyne photodynamic therapy (low or very low fluence rate) combined with intravitreal injections of bevacizumab (Avastin) compared with bevacizumab alone will, with similar safety and efficacy, delay time to retreatment with bevacizumab after the initial treatment, in subjects with new wet AMD Hypothesis: PDT in combination with Avastin at either the low or very low fluence rate will delay time to retreatment and reduce the average number of treatments required, compared to Avastin alone, but will have a similar safety and efficacy profile.

ELIGIBILITY:
Inclusion Criteria:

new wet AMD

Exclusion Criteria:

-

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2006-07; Primary Completion 2008-06 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
To determine if Visudyne therapy (low or very low fluence rate) combined with bevacizumab compared with bevacizumab alone will, with similar safety and efficacy, delay time to retreatment with bevacizumab

SECONDARY OUTCOMES:
To determine if Visudyne therapy (low or very low fluence rate) combined with bevacizumab compared with bevacizumab alone will, with similar safety and efficacy, reduce the average number of bevacizumab treatments

CONTACTS AND LOCATIONS:
Overall Officials: Michael Potter, MD, Principal Investigator — The University of British Columbia
Locations (1):
- Vancouver General Hospital Eye Care Centre (UBC), Vancouver, British Columbia, Canada